CLINICAL TRIAL: NCT02339740
Title: A Phase III Study for Patients With Newly Diagnosed Acute Promyelocytic Leukemia (APL) Using Arsenic Trioxide and All-Trans Retinoic Acid
Brief Title: Tretinoin and Arsenic Trioxide in Treating Patients With Untreated Acute Promyelocytic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAML1331; NCI-2014-02266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PAAML1331_A01PAMDREVW0; AAML1331; AAML1331 (Other: Children's Oncology Group); AAML1331 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Results first posted 2021-12-16 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Acute Promyelocytic Leukemia With t(15;17)(q24.1;q21.2); PML-RARA
MeSH Terms: interventions — Arsenic Trioxide; arsenous acid; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Idarubicin; Mitoxantrone; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (tretinoin, arsenic trioxide, chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Arsenic Trioxide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Idarubicin; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tretinoin

INTERVENTIONS:
Drug: Arsenic Trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; ATO; Trisenox; White Arsenic
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Tretinoin — Given PO
  Other Names: 2,4,6,8-Nonatetraenoic acid, 3, 7-dimethyl-9-(2,6,6-trimethyl-1-cyclohexen-1-yl)-, (all-E)-; Aberel; Airol; Aknoten; all trans-Retinoic acid; All-trans Retinoic Acid; All-trans Vitamin A Acid; all-trans-Retinoic acid; all-trans-Vitamin A acid; ATRA; Avita; beta-Retinoic Acid; Cordes Vas; Dermairol; Epi-Aberel; Eudyna; Renova; Retin-A; Retin-A MICRO; Retin-A-Micro; Retinoic Acid; Retisol-A; Ro 5488; Stieva-A; Stieva-A Forte; Trans Retinoic Acid; Trans Vitamin A Acid; trans-Retinoic Acid; Tretinoinum; Vesanoid; Vitamin A Acid; Vitamin A acid, all-trans-; Vitinoin

SUMMARY:
This phase III trial studies tretinoin and arsenic trioxide in treating patients with newly diagnosed acute promyelocytic leukemia. Standard treatment for acute promyelocytic leukemia involves high doses of a common class of chemotherapy drugs called anthracyclines, which are known to cause long-term side effects, especially to the heart. Tretinoin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Arsenic trioxide may stop the growth of cancer cells by either killing the cells, by stopping them from dividing, or by stopping them from spreading. Completely removing or reducing the amount of anthracycline chemotherapy and giving tretinoin together with arsenic trioxide may be an effective treatment for acute promyelocytic leukemia and may reduce some of the long-term side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To eliminate exposure to conventional chemotherapy (including anthracyclines), for patients with standard risk acute promyelocytic leukemia (APL), through use of arsenic trioxide (ATO) and all-trans retinoic acid (ATRA) (tretinoin) based therapy while achieving an event free survival (EFS) that is not inferior compared to historical controls.

II. To significantly reduce exposure to conventional chemotherapy, and in particular, anthracycline exposure, for patients with high risk APL, through use of ATO and ATRA based therapy while achieving an event free survival that is not inferior compared to historical controls.

EXPLORATORY OBJECTIVES:

I. To analyze the clinical impact of FMS-like tyrosine kinase 3 (FLT3) mutations in pediatric APL.

II. To correlate clinical outcomes with the kinetics of reduction in promyelocytic leukemia (PML)/retinoic acid receptor alpha (RARalpha) transcript level by quantitative real-time (RT)-polymerase chain reaction (PCR) (RQ-PCR) in bone marrow and peripheral blood samples from diagnosis to time points during therapy.

III. To monitor incidence of coagulopathy complications, utilizing standardized conventional supportive care, and correlate with a battery of coagulation testing.

IV. To evaluate the neurocognitive outcomes of patients treated on this protocol using patient-completed, performance-based measures of neuropsychological functioning and parent questionnaire report.

OUTLINE:

INDUCTION THERAPY: Patients with standard and high risk APL receive tretinoin orally (PO) twice daily (BID) and arsenic trioxide intravenously (IV) over 2-4 hours on days 1-28. High risk APL patients also receive dexamethasone PO or IV BID on days 1-14 and idarubicin IV over 15 minutes on days 1, 3, 5, and 7. Patients achieving hematologic complete remission (hCR)/hematologic complete remission with incomplete blood count recovery (hCRi) may go on to consolidation therapy. Patients who do not achieve hCR/hCRi may continue treatment with tretinoin and arsenic trioxide for up to 70 days.

CONSOLIDATION THERAPY: Patients receive tretinoin PO BID on days 1-14 and 29-42 and arsenic trioxide IV over 2-4 hours on days 1-5, 8-12, 15-19, and 22-26. Treatment repeats every 56 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then receive tretinoin PO BID on days 1-14 and arsenic trioxide IV over 2-4 hours on days 1-5, 8-12, 15-19, and 22-26.

MINIMAL RESIDUAL DISEASE (MRD) CONSOLIDATION THERAPY: Patients who have APL in the bone marrow after 2 courses of consolidation therapy receive MRD consolidation therapy prior to continuing onto consolidation course 3. Patients receive cytarabine IV over 1-3 hours every 12 hours on days 1-4; mitoxantrone hydrochloride IV over 15-30 minutes on days 3-6; and tretinoin PO BID on days 1-14. If there are no APL cells in the bone marrow after completion of MRD consolidation therapy, patients continue on to consolidation course 3.

After completion of study treatment, patients are followed up monthly for 12 months, every 3 months for 36 months, every 6 months for 48 months, and then annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with a clinical diagnosis of APL (initially by morphology of bone marrow or peripheral blood)

  * Bone marrow is highly preferred but in cases where marrow cannot be obtained at diagnosis, peripheral blood will be accepted
* If the RQ-PCR results are known at the time of study enrollment, the patient must demonstrate the PML-RARalpha transcript by RQ-PCR to be eligible
* NOTE: A lumbar puncture is not required in order to be enrolled on study nor are lumbar punctures recommended at the time of diagnosis; if the diagnosis of APL is known or suspected, diagnostic lumbar punctures in patients with neurologic symptoms should be deferred until any coagulopathy is corrected; if central nervous system (CNS) disease is suspected or proven, a computed tomography (CT) or magnetic resonance imaging (MRI) should be considered to rule out the possibility of an associated chloroma; if CNS disease is documented, patients are still eligible and will receive protocol directed intrathecal treatments
* Patients may receive up to a maximum of 5 days of pre-treatment with ATRA prior to administration of protocol therapy
* Treatment with hydroxyurea, corticosteroids (any route) and intrathecal cytarabine prior to beginning protocol directed therapy is allowed; however, it should be noted that lumbar puncture and intrathecal therapy at initial diagnosis of APL is not recommended
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with secondary APL are excluded; this includes all patients with APL that may have resulted from prior treatment (chemotherapy or radiation)
* Patients with isolated myeloid sarcoma (myeloblastoma, chloroma, including leukemia cutis) but without evidence of APL by bone marrow or peripheral blood morphology are excluded
* Patients with a pre-existing diagnosis of a prolonged QT syndrome (even if corrected QT interval [QTc] is normal at the time of APL diagnosis) are excluded
* Patients with a baseline QTc of > 450 msec are excluded; Bazett's formula is to be used for measurement of the corrected QT interval: the QT interval (msec) divided by the square root of the RR interval (msec)
* Patients with a history or presence of significant ventricular or atrial tachyarrhythmia are excluded
* Patients with right bundle branch block plus left anterior hemiblock, bifascicular block are excluded
* Patients with serum creatinine > 3.0 mg/dL and patients on active dialysis for renal dysfunction are excluded
* Patients who have received treatment with any other cytotoxic chemotherapy prior to beginning protocol therapy (other than allowed in above criteria) are excluded
* Female patients who are pregnant are excluded; patients should not be pregnant or plan to become pregnant while on treatment; a pregnancy test prior to enrollment is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants are excluded
* Sexually active patients of reproductive potential who have not agreed to be abstinent or use 2 forms of effective contraception during treatment through 1 month off therapy are excluded

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 158 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2025-09-22 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Kutny, Principal Investigator — Children's Oncology Group
Locations (174):
- United States (152):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital-Adelaide, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - Perth Children's Hospital, Perth, Western Australia
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch
- Puerto Rico (3):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Derived] Kutny MA, Alonzo TA, Abla O, Rajpurkar M, Gerbing RB, Wang YC, Hirsch BA, Raimondi S, Kahwash S, Hardy KK, Hardy S, Meshinchi S, Gamis AS, Kolb EA, Feusner JH, Gregory J Jr. Assessment of Arsenic Trioxide and All-trans Retinoic Acid for the Treatment of Pediatric Acute Promyelocytic Leukemia: A Report From the Children's Oncology Group AAML1331 Trial. JAMA Oncol. 2022 Jan 1;8(1):79-87. doi: 10.1001/jamaoncol.2021.5206. PMID 34762093
- Available data/document: Individual Participant Data Set — http://nctn-data-archive.nci.nih.gov/ — Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Risk: WBC <10,000 cells/µL
- High Risk: WBC ≥10,000 cells/µL
Period: Overall Study
Arm/Group | Standard Risk | High Risk
Started | 101 | 57
Completed | 92 | 53
Not Completed | 9 | 4
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Inevaluable-RQPCR positive not confirmed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Risk | High Risk | Total
Number analyzed (Participants) | 101 | 57 | 158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85 | 53 | 138
  Between 18 and 65 years | 16 | 4 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.9 (4.5) | 12.3 (4.7) | 13.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 25 | 73
  Male | 53 | 32 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 14 | 46
  Not Hispanic or Latino | 56 | 37 | 93
  Unknown or Not Reported | 13 | 6 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 13 | 26
  White | 60 | 34 | 94
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 18 | 7 | 25
Region of Enrollment [Number; unit: participants]
  United States | 90 | 54 | 144
  Canada | 6 | 2 | 8
  Australia | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) in Standard Risk Acute Promyelocytic Leukemia (APL) Patients
Description: EFS is defined as the time from on study to failure to achieve hematological complete response (CR) prior to start of consolidation, persistence of molecular positive disease after minimal residual disease (MRD) positive consolidation course, relapse (molecular, morphologic or extramedullary), or death. The Kaplan-Meier method will be used to estimate 2-year EFS along with 90% log-minus-log transformed confidence limits.
Time Frame: Up to 24 months
Population: Patients ineligible, did not start treatment, or RQPCR positive not confirmed are excluded from analyses of EFS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Standard Risk
Number analyzed (Participants) | 98
percentage of participants | 97.9 [93.4 to 99.3]

2. Primary Outcome: EFS in High Risk APL Patients
Description: EFS is defined as the time from on study to failure to achieve hematological CR prior to start of consolidation, persistence of molecular positive disease after MRD positive consolidation course, relapse (molecular, morphologic or extramedullary), or death. The Kaplan-Meier method will be used to estimate 2-year EFS along with 90% log-minus-log transformed confidence limits.
Time Frame: Up to 24 months
Population: Patients ineligible, did not start treatment, or RQPCR positive not confirmed are excluded from analyses of EFS
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk
Number analyzed (Participants) | 56
percentage of participants | 96.1 [88.2 to 98.8]

3. Other Pre Specified Outcome: Induction Death Rate for Patients With FLT3 Mutations and Wild Type FLT3
Description: A Fisher's exact test will be used to compare the induction death rate for patients with FLT3 mutations to patients with wild type FLT3.
Time Frame: Up to 70 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Disease Free Survival (DFS)
Description: For patients in remission at the end of induction, the log-rank test will be used to test for differences in DFS for those with end of induction real-time quantitative polymerase chain reaction (RQ-PCR) of < 1 normalized copy number (NCN) compared with those with end of Induction RQ-PCR >= 1 NCN.
Time Frame: Up to 70 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Incidence of Serious Early Coagulopathy Events, Defined as Grade 3 or Higher Hemorrhage or Thrombosis
Description: Will calculate the International Society of Thrombosis and Haemostasis (ISTH) disseminated intravascular coagulation (DIC) score and compare the sensitivity and specificity of ISTH with that of thrombomodulin using McNemar's test for paired data. To improve the predictive ability of the ISTH DIC score, will use a stepwise combination of biomarkers. Receiver operating characteristic (ROC) curve will be used to assess the accuracy in prediction of bleeding events during induction and the areas under the ROC curve will be compared.
Time Frame: Up to 29 days of induction therapy
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in CogState Scores, Defined as a Decline of 5 Units in Mean Scores Apparent at 2 Years Off Therapy
Description: Actual CogState scores for each domain at each time point will be summarized and examined by descriptive statistics and scatter plots. Change in score for a domain from end of induction will be calculated and summarized by descriptive statistics. The mean change of score from end of induction to a later time-point will be estimated with its 95% confidence interval. Linear mixed models using scores from all time-points as outcome will also be used to estimate the change in scores between time-points with adjustment for within-patient correlation of the score by random effects for individual patients.
Time Frame: End of induction up to 2 years post-treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Parent-reported Executive Functioning Over Time, Defined as a Decline of 5 Units in Mean Scores Apparent at 2 Years Off Therapy
Description: Measured by the Behavioral Regulation, Working Memory and Metacognition Indices of the Behavior Rating Inventory of Executive Function. Change in score for a domain from end of induction will be calculated and summarized by descriptive statistics. The mean change of score from end of induction to a later time-point will be estimated with its 95% confidence interval. Linear mixed models using scores from all time-points as outcome will be used to estimate change in scores between time-points with adjustment for within-patient correlation of the score by random effects for individual patients.
Time Frame: End of induction up to 2 years post-treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Intellectual Functioning, Defined by Declines on the Wechsler-derived Estimated Intelligence Quotient and Processing Speed Scores
Description: One sample t-test on the change of score will be used to examine if there is significant decline in neurocognitive function from end of induction to 2 years off therapy. Linear mixed models using scores from all time-points as outcome will also be used to estimate the change in scores between time-points with adjustment for within-patient correlation of the score by random effects for individual patients.
Time Frame: End of treatment to 4 years post-treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Memory Functioning, Defined by Declines on the Children's Memory Scale Faces and Stories Memory Scores
Description: as for outcome 8
Time Frame: End of treatment to 4 years post-treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Verbal Learning Functioning, Defined by Declines on the California Verbal Learning Test Total Score
Description: as for outcome 8
Time Frame: End of treatment to 4 years post-treatment
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Adaptive Functioning, Defined by Declines on the Adaptive Behavior Assessment System-II General Adaptive Behavior Composite Score
Description: as for outcome 8
Time Frame: End of treatment to 4 years post-treatment
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Parent-reported Psychosocial Functioning Over Time
Description: Psychosocial functioning over time as defined by declines on the Behavior Assessment System for Children-Second Edition (BASC-2) Anxiety, Depression, and Social Skills scores, and the Pediatric Quality of Life Inventory (PedsQL) Total and Physical Health scores.
Time Frame: End of treatment to 4 years off-therapy
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Parent-reported Quality of Life (QOL) Over Time
Description: QOL over time as defined as declines on the BASC-2 Anxiety, Depression, and Social Skills scores, and the PedsQL Total and Physical Health scores.
Time Frame: End of treatment to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on protocol therapy (including up to 6 courses) or during follow-up.
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Standard Risk | High Risk
All-Cause Mortality (participants affected / at risk) | 1/101 | 0/57
Serious Adverse Events (participants affected / at risk) | 3/101 | 2/57
Other Adverse Events (participants affected / at risk) | 89/101 | 50/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Risk (N=101) | High Risk (N=57)
Death NOS (General disorders) | 1 | 0 (0)
Multi-organ failure (General disorders) | 1 | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 | 0 (0)
Encephalopathy (Nervous system disorders) | 1 | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 (0)
Seizure (Nervous system disorders) | 1 | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Risk (N=101) | High Risk (N=57)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 4 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Papilledema (Eye disorders) | 3 | 1
Periorbital edema (Eye disorders) | 1 | 0
Vitreous hemorrhage (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 11
Nausea (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Fever (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 1
Bone infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 3 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 7 | 5
Kidney infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 16 | 6
Aspartate aminotransferase increased (Investigations) | 11 | 4
Blood bilirubin increased (Investigations) | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 67 | 43
Fibrinogen decreased (Investigations) | 1 | 6
Investigations - Other, specify (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 0
Weight gain (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 4
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 8 | 4
Intracranial hemorrhage (Nervous system disorders) | 0 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 2 | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 2
Hematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 4 | 2
Thromboembolic event (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT02339740/Prot_SAP_000.pdf